CLINICAL TRIAL: NCT05455671
Title: Real-Time Assessment of Lung Structure and Function in Children and Young Adults With CF Using Electrical Impedance Tomography
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0114
Record Dates: First submitted 2022-06-06; First posted 2022-07-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis; Healthy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 - Healthy Controls: Persons, male or female, between the ages of 3 and 21 (inclusive) with healthy lungs, defined by no known or suspected chronic or temporary lung disease. A single study visit
- Cohort 2 - CF Longitudinal: Persons, male or female, with CF, defined by two known disease-causing mutations and/or a sweat chloride value of >60mmol/L, between the ages of 3 and 21 (inclusive).
- Cohort 3 - CF Exacerbation: Persons, male or female, with CF, defined by two known disease-causing mutations and/or a sweat chloride value of >60mmol/L, between the ages of 3 and 21 (inclusive), experiencing a pulmonary exacerbation requiring antibiotics.

SUMMARY:
The purpose of this study is to determine the ability of electrical impedance tomography (EIT) to identify structural and functional physiological changes that occur with disease progression in cystic fibrosis patients. The investigators also aim to determine whether EIT can serve as an alternative for CT to identify regions of air trapping and consolidation, whether EIT can provide clinically useful information about response to treatment for an acute PE, and whether EIT can provide longitudinal information about structural changes in the lung.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Age 3-21 years
* Male or female
* Healthy subjects with no known or suspected chronic or temporary lung disease

Cohort 2:

* Age 3-21 years
* Male or female
* CF as diagnosed based on sweat chloride value(>60 mmol/L) or two known disease causing mutations

Cohort 3:

* Age 3-21 years
* Male or female
* CF as diagnosed based on sweat chloride value (>60 mmol/L) or two known disease causing mutations
* Experiencing a protocol defined pulmonary exacerbation and being started on oral or intravenous antibiotics

Exclusion Criteria:

* Unwilling/refusal to sign consent
* Known congenital heart disease, arrhythmia, or history of heart failure
* Wearing a pacemaker or a metallic surgical implant in the chest
* History of infection with Burkholderia cepacia
* Developmental delays that could result in an inability to complete study procedures

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and young adults between 3 and 21 years old, with or without cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Identification of air trapping and consolidation by EIT | 36 months
  The detection task for identifying air trapping and consolidation is to determine by inspection regions of EIT VQ index significantly lower than the surrounding lung region, with actual numbers or relative differences to be determined as part of this study in the correlation analysis to CT scans.

SECONDARY OUTCOMES:
Determining utility of EIT information in response to treatment for a pulmonary exacerbation | 36 months
  Individual outcome measures (CFCS, LCI , PFT, and EIT measures) will be evaluated using paired t-tests, and the corresponding t-statistics from each of the tests will be used as measures of effect size for comparison. In addition, all of the clinical outcomes can be compared statistically using a joint model approach (this is the same model that is referenced in Q3 below).
Determination of structural changes in the lung by EIT | 36 months
  The EIT-derived global VQ indices, FEV1, FEV1/FVC, FVC, and extent of air trapping and consolidation will be studied longitudinally and compared to LCIs, PFTs, and CT scans when available to assess the ability of EIT to identify structural and reversible physiological changes that occur with disease progression. To estimate the change in the EIT measures of global VQ, air trapping and consolidation, and EIT-derived PFT outputs over time, a random coefficient model with an intercept and slope fit for each subject with at least two measurements over the 3 years will be used. A bivariate version of the random coefficients model will be fit to address whether the EIT outcome variable is associated with the spirometer PFT outputs, LCI, and CFCS while accounting for repeated measures.

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Jordana, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No